CLINICAL TRIAL: NCT00799396
Title: Pharmacogenomics of Anti-Platelet Interventions (The PAPI Study)
Brief Title: Determining Genetic Role in Treatment Response to Anti-Platelet Interventions (The PAPI Study)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Alan Shuldiner, Associate Dean for Personalized Medicine; Director, Program in Personalized and Genomic Medicine; Head, Division of Endocrinology, Diabetes and Nutrition, University of Maryland, Baltimore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HP-00043419; U01 HL074518-01; U01GM074518 (NIH)
Record Dates: First submitted 2008-11-26; First posted 2008-11-27 (Estimated); Results first posted 2016-03-28 (Estimated); Last update posted 2022-02-24 (Actual); Status verified 2022-02

CONDITIONS: Platelet Aggregation Inhibitors; Coronary Heart Disease
MeSH Terms: conditions — Coronary Disease | interventions — Clopidogrel; Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Overall Study (Experimental): Participants will receive clopidogrel treatment alone, followed by clopidogrel plus aspirin treatment on the last day of treatment.
  Interventions: Drug: Clopidogrel; Drug: Aspirin

INTERVENTIONS:
Drug: Clopidogrel — 300 mg on first day, then 75 mg per day for the next 6 days
Drug: Aspirin — Single dose of 324 mg on the last day of clopidogrel treatment

SUMMARY:
One of the most common ways for preventing coronary heart disease (CHD) is to take aspirin or clopidogrel. However, studies have shown that not all people respond to these medications. The variance in treatment response may be linked to genetics. This study will examine the effects of aspirin and clopidogrel in a population whose genes are well known in order to determine the role that genes play in treatment responses.

DETAILED DESCRIPTION:
CHD is the leading cause of death in the United States. Anti-platelet agents lessen platelet aggregation and are used commonly to prevent recurrent CHD events. Two of the most common anti-platelet agents are aspirin and clopidogrel. However, up to 25% to 30% of people do not respond to these medications. Evidence indicates that treatment response may be related to genetics. The purpose of this study is to determine specific gene variants that predict response to aspirin and clopidogrel therapy.

This study is part of a larger group of studies called the Pharmacogenomics Research Network (PGRN). Participants will include the Old Order Amish of Lancaster, Pennsylvania. They are well suited for genetic studies because they are a homogenous, closed, founder population. Participants will receive 300 mg of clopidogrel on the first day, then 75 mg of clopidogrel per day for the next 6 days. On the last day of clopidogrel treatment, participants will take a single dose of 324 mg aspirin. Participants will undergo platelet function tests before and after clopidogrel alone, and then again after taking clopidogrel plus aspirin. Using the gene variation profiles across the genome, researchers will analyze which genes correspond to treatment response.

ELIGIBILITY:
Inclusion Criteria:

* Of Old Order Amish descent

Exclusion Criteria:

* Currently pregnant or less than 6 months have passed since delivery
* Has a history of a bleeding disorder or major spontaneous bleed, such as peptic ulcer, epistasis, or intracranial bleed
* Has severe hypertension, defined by a blood pressure above 160/95 mm Hg, making it unethical not to recommend prompt treatment
* Takes medications that would affect the outcome(s) to be measured and cannot willingly and safely, in the opinion of the treating physician and study physician, discontinue these medications for 1 week prior to protocol initiation
* Is taking vitamins or other supplements and is unwilling to discontinue their use for at least 1 week prior to study
* Has a coexisting malignancy
* Has a creatinine level greater than 2.0 mg/dl, aspartate transaminase (AST) or alanine transaminase (ALT) greater than two times the upper limit of normal, hematocrit less than 32%, or a thyroid-stimulating hormone (TSH) less than 0.4 or greater than 5.5 mIU/L
* Has a bleeding disorder or history of gastrointestinal bleeding or other major bleeding episode
* Is currently taking aspirin, clopidogrel, or other anti-coagulant, such as warfarin, heparin, or GPIIb/IIIa antagonists, and have conditions that might place them at increased risk from withdrawal of these medications 14 days prior to protocol initiation, including history of unstable angina, heart attack, angioplasty (including stent placement), coronary artery bypass surgery, atrial fibrillation, stroke or transient ischemic attacks, diabetes, or deep vein thrombosis or other thrombosis
* Has polycythemia, or thrombocytosis, defined by a platelet count greater than 500,000
* Has thrombocytopenia, defined by a platelet count less than 75,000
* Has had surgery within the last 6 months
* Has an aspirin or clopidogrel allergy
* Currently breast feeding

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 682 (Actual)
Dates: Start 2006-07; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan R. Shuldiner, MD, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- Amish Research Clinic, Lancaster, Pennsylvania, United States

REFERENCES:
- [Result] Shuldiner AR, O'Connell JR, Bliden KP, Gandhi A, Ryan K, Horenstein RB, Damcott CM, Pakyz R, Tantry US, Gibson Q, Pollin TI, Post W, Parsa A, Mitchell BD, Faraday N, Herzog W, Gurbel PA. Association of cytochrome P450 2C19 genotype with the antiplatelet effect and clinical efficacy of clopidogrel therapy. JAMA. 2009 Aug 26;302(8):849-57. doi: 10.1001/jama.2009.1232. PMID 19706858
- [Result] Bozzi LM, Mitchell BD, Lewis JP, Ryan KA, Herzog WR, O'Connell JR, Horenstein RB, Shuldiner AR, Yerges-Armstrong LM. The Pharmacogenomics of Anti-Platelet Intervention (PAPI) Study: Variation in Platelet Response to Clopidogrel and Aspirin. Curr Vasc Pharmacol. 2016;14(1):116-24. doi: 10.2174/1570161113666150916094829. PMID 26374108
- [Result] Lewis JP, Ryan K, O'Connell JR, Horenstein RB, Damcott CM, Gibson Q, Pollin TI, Mitchell BD, Beitelshees AL, Pakzy R, Tanner K, Parsa A, Tantry US, Bliden KP, Post WS, Faraday N, Herzog W, Gong Y, Pepine CJ, Johnson JA, Gurbel PA, Shuldiner AR. Genetic variation in PEAR1 is associated with platelet aggregation and cardiovascular outcomes. Circ Cardiovasc Genet. 2013 Apr;6(2):184-92. doi: 10.1161/CIRCGENETICS.111.964627. Epub 2013 Feb 7. PMID 23392654
- [Result] Lewis JP, Horenstein RB, Ryan K, O'Connell JR, Gibson Q, Mitchell BD, Tanner K, Chai S, Bliden KP, Tantry US, Peer CJ, Figg WD, Spencer SD, Pacanowski MA, Gurbel PA, Shuldiner AR. The functional G143E variant of carboxylesterase 1 is associated with increased clopidogrel active metabolite levels and greater clopidogrel response. Pharmacogenet Genomics. 2013 Jan;23(1):1-8. doi: 10.1097/FPC.0b013e32835aa8a2. PMID 23111421
- [Result] Lewis JP, Fisch AS, Ryan K, O'Connell JR, Gibson Q, Mitchell BD, Shen H, Tanner K, Horenstein RB, Pakzy R, Tantry US, Bliden KP, Gurbel PA, Shuldiner AR. Paraoxonase 1 (PON1) gene variants are not associated with clopidogrel response. Clin Pharmacol Ther. 2011 Oct;90(4):568-74. doi: 10.1038/clpt.2011.194. Epub 2011 Aug 31. PMID 21881565
- [Result] Lewis JP, Stephens SH, Horenstein RB, O'Connell JR, Ryan K, Peer CJ, Figg WD, Spencer SD, Pacanowski MA, Mitchell BD, Shuldiner AR. The CYP2C19*17 variant is not independently associated with clopidogrel response. J Thromb Haemost. 2013 Sep;11(9):1640-6. doi: 10.1111/jth.12342. PMID 23809542
- [Derived] Bergmeijer TO, Reny JL, Pakyz RE, Gong L, Lewis JP, Kim EY, Aradi D, Fernandez-Cadenas I, Horenstein RB, Lee MTM, Whaley RM, Montaner J, Gensini GF, Cleator JH, Chang K, Holmvang L, Hochholzer W, Roden DM, Winter S, Altman RB, Alexopoulos D, Kim HS, Dery JP, Gawaz M, Bliden K, Valgimigli M, Marcucci R, Campo G, Schaeffeler E, Dridi NP, Wen MS, Shin JG, Simon T, Fontana P, Giusti B, Geisler T, Kubo M, Trenk D, Siller-Matula JM, Ten Berg JM, Gurbel PA, Hulot JS, Mitchell BD, Schwab M, Ritchie MD, Klein TE, Shuldiner AR; ICPC Investigators. Genome-wide and candidate gene approaches of clopidogrel efficacy using pharmacodynamic and clinical end points-Rationale and design of the International Clopidogrel Pharmacogenomics Consortium (ICPC). Am Heart J. 2018 Apr;198:152-159. doi: 10.1016/j.ahj.2017.12.010. Epub 2017 Dec 17. PMID 29653637
- [Derived] Salimi S, Lewis JP, Yerges-Armstrong LM, Mitchell BD, Saeed F, O'Connell JR, Perry JA, Ryan KA, Shuldiner AR, Parsa A. Clopidogrel Improves Skin Microcirculatory Endothelial Function in Persons With Heightened Platelet Aggregation. J Am Heart Assoc. 2016 Oct 31;5(11):e003751. doi: 10.1161/JAHA.116.003751. PMID 27799230
- See also: dbGaP submission for the PAPI study — http://www.ncbi.nlm.nih.gov/projects/gap/cgi-bin/study.cgi?study_id=phs000391.v1.p1

RESULTS

PARTICIPANT FLOW:
Period: Clopidogrel Treatment
Arm/Group | Overall Study
Started | 682
Completed | 669
Not Completed | 13
Not completed — Adverse Event | 6
Not completed — Physician Decision | 5
Not completed — Withdrawal by Subject | 2
Period: Clopidogrel Plus Aspirin
Arm/Group | Overall Study
Started | 669
Completed | 663
Not Completed | 6
Not completed — Adverse Event | 2
Not completed — Physician Decision | 4

BASELINE CHARACTERISTICS:
Population: Participants were recruited from the Old Order Amish of Lancaster, Pennsylvania. They are well suited for genetic studies because they are a homogenous, closed, founder population.
Arm/Group | Overall Study
Number analyzed (Participants) | 682
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.5 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 343
  Male | 339
Region of Enrollment [Number; unit: participants]
  United States | 682

OUTCOME MEASURES:

1. Primary Outcome: Changes in Platelet Function in Response to Clopidogrel
Description: Baseline minus post clopidogrel/pre-aspirin platelet rich plasma (PRP) maximum aggregation.
Time Frame: Measured at baseline, and after clopidogrel treatment
Measure: Mean (Standard Deviation); unit: percentage of maximum aggregation change
Groups:
- Overall Study: Participants will receive clopidogrel treatment alone, followed by clopidogrel plus aspirin treatment on the last day of treatment.
  Clopidogrel: 300 mg on first day, then 75 mg per day for the next 6 days
  Aspirin: Single dose of 324 mg on the last day of clopidogrel treatment
  PRP ADP 20 = Platelet Rich Plasma ADP-induced (20 microM) aggregation
  PRP Collagen 5 = Platelet Rich Plasma Collegan-induced (5 microM) aggregation
Arm/Group | Overall Study
Number analyzed (Participants) | 669
percentage of maximum aggregation change
  PRP ADP 20 | 38.51 (14.30)
  PRP Collagen 5 | 14.06 (15.01)

2. Primary Outcome: Changes in Platelet Function in Response to Clopidogrel Plus Aspirin
Description: Baseline minus post clopidogrel/post-aspirin platelet rich plasma (PRP) maximum aggregation
Time Frame: Measured at baseline, and after clopidogrel plus aspirin treatment
Measure: Mean (Standard Deviation); unit: percentage of max aggregation change
Arm/Group | Overall Study
Number analyzed (Participants) | 663
percentage of max aggregation change
  PRP ADP 20 | 41.21 (13.09)
  PRP Collagen 5 | 56.64 (14.44)

ADVERSE EVENTS:
Time Frame: 37 days
Description: Adverse event data were collected during both intervention periods and for 30 days after the final study visit. There were 6 Adverse Events during the Clopidogrel Treatment Arm and 2 Adverse Events during the Clopidogrel plus Aspirin Arm. This does not exceed the threshold for reporting Other Adverse Events.
Arm/Group | Overall Study
Serious Adverse Events (participants affected / at risk) | 0/682
Other Adverse Events (participants affected / at risk) | 0/682

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes